CLINICAL TRIAL: NCT00922597
Title: Non-interventional Observation of Practical Implementation, Efficacy and Safety of Continuous Infusion With KOGENATE Bayer in Surgery - NO PEACKS
Brief Title: Non-interventional Observation of Practical Implementation, Efficacy and Safety of Continuous Infusion With KOGENATE Bayer in Surgery
Acronym: NO PEACKS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13213; KG0701 (Other: Company internal)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Hemophilia A
Keywords: Continuous infusion; Surgery; Severe haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Patients undergoing surgery and receiving continuous infusion with Kogenate Bayer according to local drug information.

SUMMARY:
The objective of this international post-marketing surveillance study is to collect data on the efficacy and safety of continuous infusion with KOGENATE Bayer in surgery.

ELIGIBILITY:
Inclusion Criteria:

* In-patients with diagnosis of severe haemophilia A (FVIII < 1%), heavily pretreated (> 150 exposure days), without any history of inhibitors, a negative inhibitor test should be available, decision taken by the investigator to administer KOGENATE Bayer via continuous infusion during and after surgery.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of severe haemophilia A. Physicians should consult the full prescribing information for KOGENATE Bayer before enrolling patients and familiarize themselves with the safety information in the product information.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-08; Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Total consumption of FVIII (in IU/kg) during continuous infusion, FVIII:C achieved compared to expected levels, reasons and number of unplanned bolus infusion, amount of blood loss, transfusion requirements | During continuous infusion

SECONDARY OUTCOMES:
General tolerability and development of inhibitors | Within 14 days to 3 months after termination of continuous infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Many Locations, Austria
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Italy
- Many Locations, Netherlands
- Many Locations, Slovenia
- Many Locations, Spain